CLINICAL TRIAL: NCT05221372
Title: proSpecTive sAmpling in dRiver muTation Pulmonary Oncology Patients on Tyrosine Kinase Inhibitors
Brief Title: ProSpecTive sAmpling in dRiver muTation Pulmonary Oncology Patients on Tyrosine Kinase Inhibitors (START-TKI)
Acronym: START-TKI
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Anne-Marie Dingemans, MD, PhD, Erasmus Medical Center
Other Study IDs: NL58664.078.16
Record Dates: First submitted 2022-01-10; First posted 2022-02-03 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Non Small Cell Lung Cancer; Liquid Biopsy; Tyrosine Kinase Inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Circulating tumor DNA on blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is perfomed with adult patients with non-small cell lung cancer treated with tyrosine kinase inhibitor. The objective is to collect repeated samples of blood from patients (starting) on a tyrosine kinase inhibitor, for liquid mutation testing, and pharmacokinetic analysis.

DETAILED DESCRIPTION:
This is an observational study in pulmonary oncology patients treated with TKI. Ideally before start of therapy, at week 4, 8 12, and then every 4-8 weeks (following the standard of care clinical pathways local guidelines) extra tubes of blood will be collected during blood withdrawal planned for standard-of-care. When a TKI switch takes place, patients receive a new study number and the blood collection will be continued following standard-of-care. Sampling will be performed during steady-state in working hours before next ingestion of TKI (the regular morning dose will need to be postponed until after blood withdrawal).

The moment of blood withdrawal after start of therapy and after last dosage of TKI will be registered.

At the time of progression the current standard of care is to perform a rebiopsy, to identify the resistance mechanism and determine the next appropriate systemic therapy for a patient. Some mechanisms can only be determined on a biopsy specimen (e.g. transformation to SCLC, MET amplification FISH). This study is observational and will not interfere with the current standard practice, therefore the treating physician is free to determine the indication for and possibility of a rebiopsy. However, when a biopsy is taken as standard of care, we will also draw an extra blood sample on the day of the biopsy (preferably during standard preprocedural coagulation status laboratory investigations) and use a portion of the biopsy for a fresh frozen specimen, as evolving molecular investigations (like RNA analysis) often need fresh non-fixed material to obtain reliable results.

Four to five core biopsies will be obtained for further analysis. Half of the obtained biopsy material will be stored in formalin according to local standard procedures, while the other half will be fresh frozen according to local standard procedures and stored for further analysis.

When the treating physician needs to take additional tissue or liquid (e.g. pleural fluid, liquor) for investigations following standard-of-care protocols, we would like to perform additional molecular and/or pharmacokinetic analysis on the residual material when applicable.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Able to understand the written informed and able to give informed consent
* Locally advanced or metastatic NSCLC with oncogenic driver mutation
* Treatment with TKI according to standard of care

Exclusion Criteria:

* Unable to draw blood for study purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with non-small cell lung cancer treated with a tyrosine kinase inhibitor
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2017-02-02 (Actual); Primary Completion 2031-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Relative presence of primary mutation and resistance mutations in plasma levels under treatment of a small molecule kinase inhibitor until progression of disease measured in variant allele frequency | 10 years
  Describing the plasma levels of primary mutations and resistance mutations under treatment by sequentially measuring cell free tumor DNA.
  Different techniques will be used for the plasma mutation detection (ddPCR and NGS)
Plasma concentrations of the small molecule kinase inhibitor during treatment until progression of disease | 10 years
  Describing the plasma concentrations over time during treatment with a small molecule kinase inhibitor by sequentially measuring mean concentrations of the small molecule kinase inhibitor.

SECONDARY OUTCOMES:
Time to progression or death under treatment with small molecule kinase inhibitor | 10 years
  Time to progression or death is defined as time from start of the small molecule kinase inhibitor to radiological progression (according to measurements conform RECIST v.1.1) or death.
Overall survival | 10 years
  Defined as time from start of the small molecule kinase inhibitor to death.
Pharmacokinetics of intratumoral small molecule kinase inhibitors | 10 years
  Measuring intratumoral concentrations of small molecule kinase inhibitors on tumor biopsy taken as part of regular care
Correlation of mutation status in blood to (re)biopsy specimen results performed for standard-of-care. | 10 years
  Concordance of detection of tumor mutations will be evaluated between ddPCR, NGS in blood, and NGS in tissue samples when available
Correlation between the BMI of the patient and mean concentration of the small molecule kinase inhibitor | 10 years
  Effects of BMI on PK will be explored by means of regression analysis.
Correlation between smoking status of the patients and mean concentration of the small molecule kinase inhibitor | 10 years
  Effects of smoking status on PK will be explored by means of regression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie Dingemans, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Steendam CMJ, Veerman GDM, Pruis MA, Atmodimedjo P, Paats MS, van der Leest C, von der Thusen JH, Yick DCY, Oomen-de Hoop E, Koolen SLW, Dinjens WNM, van Schaik RHN, Mathijssen RHJ, Aerts JGJV, Dubbink HJ, Dingemans AC. Plasma Predictive Features in Treating EGFR-Mutated Non-Small Cell Lung Cancer. Cancers (Basel). 2020 Oct 29;12(11):3179. doi: 10.3390/cancers12113179. PMID 33138052
- [Derived] Ernst SM, Uzun S, Paats MS, van Marion R, Atmodimedjo PN, de Jonge E, van Schaik RHN, Aerts JGJV, von der Thusen JH, Dubbink HJ, Dingemans AC. Efficacy and Tolerability of Osimertinib and Sotorasib Combination Treatment for Osimertinib Resistance Caused by KRAS G12C Mutation: A Report of Two Cases. JCO Precis Oncol. 2023 Sep;7:e2300451. doi: 10.1200/PO.23.00451. PMID 38096473

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT05221372/Prot_SAP_000.pdf